CLINICAL TRIAL: NCT03840759
Title: A Pilot Study of the Short-term Effects of an Inpatient Geriatric Consultation Team on Geriatric Syndrome Patients
Brief Title: Short-term Effects of an Inpatient Geriatric Consultation Team on Geriatric Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG8F1571
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2016-12

CONDITIONS: Depression; Senile Dementia
MeSH Terms: conditions — Depression; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- usual care (Experimental): For the intervention group, a geriatric physician was consulted and recommendations were made by the geriatric consultant and inpatient geriatric consultation team after a complete geriatric assessment (CGA). The CGA includes the assessment of depression, dementia, physical performance of Activity of Daily Living (ADL) and nutrition using Geriatric Depression Scale (GDC-15), Mini-Mental State Examination (MMSE), Barthel Index (BI), and Mini Nutritional Assessment-Short Form (MNA®-SF) respectively. Besides the geriatric physician, our multidisciplinary team included a social worker, nutritionist and physical therapist. In the control group, the participants only received routine hospital care and no geriatric physician was consulted.
  Interventions: Other: inpatient geriatric consultation team

INTERVENTIONS:
Other: inpatient geriatric consultation team — For the intervention group, a geriatric physician was consulted and recommendations were made by the geriatric consultant after a complete CGA.

SUMMARY:
Patients admitted to acute ordinary wards in a medical center in Southern Taiwan from an elder-integrated outpatient department or emergency room from January 2017 to December 2017 were included if they met the following criteria: (i) age 65 years or older, (ii) Barthel index score ≦60 and (iii) with at least one of the following geriatric syndromes: unsteady gait or easy-to-fall ( falls ≧ 2 in last 1 year), malnutrition with Mini Nutritional Assessment-Short Form screening score < 12, urinary incontinence, pressure sores, dementia, delirium, depression, polypharmacy (≧8 medications), and excessive utilization of healthcare facilities (admission≧2, visit Emergency≧2, or visit outpatient department≧12 in one month). Patients were excluded if they were in a vegetative state, under palliative care or terminally ill and suffering from acute illness needing to be transferred to or cared for in the Intensive Care Unit.

Human participant approval was obtained from the Chang Gung Medical Foundation Institutional Review Board before data collection. Participants were recruited from the ordinary wards by research assistants who screened the admission list every morning if they met the inclusion criteria. Then, the detail of the research was explained to the patients and families. They were allowed to choose to be in the control group or the intervention group. After the participants and or family agreed, informed consent was signed. For those who were cognitively impaired or suffered from dementia, informed consent was signed by their relative or partner. For the intervention group, a geriatric physician was consulted and recommendations were made by the geriatric consultant after a complete geriatric assessment. Besides the geriatric physician, the investigator's multidisciplinary team included a social worker, nutritionist and physical therapist. In the control group, the participants only received routine hospital care and no geriatric physician was consulted.

DETAILED DESCRIPTION:
Participants were recruited from the ordinary wards by research assistants who screened the admission list every morning if they met the inclusion criteria. Then, the detail of the research was explained to the patients and families. They were allowed to choose to be in the control group or the intervention group. After the participants and or family agreed, informed consent was signed. For those who were cognitively impaired or suffered from dementia, informed consent was signed by their relative or partner. For the intervention group, a geriatric physician was consulted and recommendations were made by the geriatric consultant after a complete CGA. The CGA includes the assessment of depression, dementia, physical performance of Activity of Daily Living (ADL) and nutrition using Geriatric Depression Scale (GDC-15), Mini-Mental State Examination (MMSE), Barthel Index (BI), and Mini Nutritional Assessment-Short Form (MNA®-SF) respectively. Besides the geriatric physician, our multidisciplinary team included a social worker, nutritionist and physical therapist. In the control group, the participants only received routine hospital care and no geriatric physician was consulted. The case manager nurse filed the participant's baseline data and clinical problems. After discharge, the participant's condition was assessed via telephone in the first, third and six months after discharge.

ELIGIBILITY:
Inclusion Criteria:

(i) age 65 years or older, (ii) Barthel index (BI) [18] score ≦60 and (iii) with at least one of the following geriatric syndromes: unsteady gait or easy-to-fall ( falls ≧ 2 in last 1 year), malnutrition with Mini Nutritional Assessment-Short Form (MNA®-SF) screening score < 12, urinary incontinence, pressure sores, dementia, delirium, depression, polypharmacy (≧8 medications), and excessive utilization of healthcare facilities (admission≧2, visit Emergency≧2, or visit outpatient department≧12 in one month)-

Exclusion Criteria:

Patients were excluded if they were in a vegetative state, under palliative care or terminally ill and suffering from acute illness needing to be transferred to or cared for in the Intensive Care Unit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
readmission rate | readmission rate within one month after discharge
  compare the differences of readmission rates between the intervention and control groups
readmission rate | readmission rate within three months after discharge
  compare the differences of readmission rates between the intervention and control groups
readmission rate | readmission rate within six months after discharge
  compare the differences of readmission rates between the intervention and control groups

SECONDARY OUTCOMES:
mortality rate | mortality rate within one month after discharge
  compare the differences of mortality rates between the intervention and control groups
mortality rate | mortality rate within three months after discharge
  compare the differences of mortality rates between the intervention and control groups
mortality rate | mortality rate within six months after discharge
  compare the differences of mortality rates between the intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Song-Seng Loke, Study Director

IPD SHARING:
Plan to Share IPD: No